CLINICAL TRIAL: NCT04223648
Title: A Pilot Study Using Programmed Cell Death 1 + Selected Cell Therapy With Durvalumab (MEDI4736) and Tremelimumab in Metastatic Melanoma
Brief Title: Programmed Cell Death 1 + Selected Cell Therapy With Durvalumab (MEDI4736) and Tremelimumab in Metastatic Melanoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Yale University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025925
Record Dates: First submitted 2019-12-19; First posted 2020-01-10 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Subjects will receive 1 cycle of tremelimumab/durvalumab
  * Subjects will undergo resection to obtain tumor for generation of autologous tumor infiltrating lymphocytes (TIL) cultures and blood draw to obtain peripheral blood mononuclear cell (PBMC)s
  * TIL and PBMC will undergo immunoselection based on binding to an anti-programmed cell death 1 (PD-1) antibody and then will be expanded ex vivo.
  Subjects will receive 3 cycles of ipilimumab/nivolumab
  • Subjects will undergo staging with computer tomography (CT) chest/abdomen/pelvis and brain magnetic resonance imaging (MRI) or CT scan.
  subjects with stable disease will continue with nivolumab monotherapy; Subjects with progressive disease will proceed to cell therapy.
  Interventions: Drug: tremelimumab/durvalumab, ipilimumab/nivolumab and nivolumab monotherapy

INTERVENTIONS:
Drug: tremelimumab/durvalumab, ipilimumab/nivolumab and nivolumab monotherapy — Subjects will receive 1 cycle of tremelimumab/durvalumab
  * Subjects will undergo resection to obtain tumor for generation of autologous tumor infiltrating lymphocytes (TIL) cultures and blood draw to obtain peripheral blood mononuclear cell (PBMC)s
  * TIL and PBMC will undergo immunoselection based on binding to an anti-programmed cell death 1 (PD-1) antibody and then will be expanded ex vivo.
  Subjects will receive 3 cycles of ipilimumab/nivolumab
  • Subjects will undergo staging with computer tomography (CT) chest/abdomen/pelvis and brain magnetic resonance imaging (MRI) or CT scan.
  subjects with stable disease will continue with nivolumab monotherapy; Subjects with progressive disease will proceed to cell therapy.

SUMMARY:
The primary objective of this pilot study is to assess the feasibility of mobilizing PD-1+ T cells to the peripheral blood after a single treatment with tremelimumab/durvalumab in patients with treatment naïve metastatic melanoma.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to assess the feasibility of mobilizing programmed cell death (PD-1)+ T cells to the peripheral blood after a single treatment with tremelimumab/durvalumab in patients with treatment naïve metastatic melanoma.

Secondary objectives are to evaluate the safety and clinical activity of administering a regimen of PD-1+ selected tumor infiltrating lymphocytes (TIL)/(Interleukin) IL-2, using a cell product manufactured in the Yale Advanced Cell Therapy Laboratories and assess for clinical activities in subjects with metastatic melanoma who are not responding or have progressed after receiving first-line therapy with 1 cycle of tremelimumab/durvalumab followed by 3 cycles of ipilimumab/nivolumab followed by nivolumab monotherapy as maintenance treatment.

Exploratory objective are to:

1. assess the number of PD-1+ T cells in the tumor microenvironment before and after a single treatment with tremelimumab/durvalumab.
2. conduct a preliminary assessment of the TCR clonotypes present in PD1+ cluster of differentiation 8 (CD8)+ cells (4-1BB, LAG-3, TIM-3, PD-1) versus PD1-CD8+ T-cells early in the expansion cultures and compare to clonotypes late in the final product and in peripheral blood lymphocytes (PBL) 1 and 2 months post infusion.
3. assess neoantigens present in resected tumor and correlate T cell specificity for neoantigens from TIL and peripheral blood mononuclear cell (PBMC) populations stratified by PD-1 expression in these cell populations.

ELIGIBILITY:
Inclusion Criteria:

Untreated metastatic melanoma

* A metastatic lesion at least 1.5 cm in diameter that can be removed surgically
* Measurable or evaluable disease not including the resected lesion; at least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to enrollment
* Capable of giving signed informed consent
* Age >18 years at time of screening
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Body weight >30 kg
* Hemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC ≥1.0 x 109/L (> 1000 per mm3)
* Absolute lymphocyte count (ALC ≥0.5 x 109/L (> 500 per mm3) Platelet count ≥100 (or 75) x 109/L (>75,000 per mm3)
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome)
* Aspartate aminotransferase (AST) (SGOT)/Alanine aminotransferase (ALT) (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

Received prior treatment for metastatic melanoma

* Received prior cell transfer therapy that included non-myeloablative or ablative chemotherapy
* Received anti PD-1 immune therapy within prior 6 months
* Any contraindication to neutropenia or thrombocytopenia for up to 2 weeks (no active major infection, no site of active, clinically significant bleeding)
* Concurrent major medical illnesses
* Any form of immunodeficiency
* Severe hypersensitivity to any of the agents used in this study
* Contraindications for IL-2 administration
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab, tremelimumab, ipilimumab or nivolumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (HBV) (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
PD1+ cell pharmacodynamic response in blood to tremelimumab/durvalumab treatment | up to 10 days post-enrollment.
  PD response is achieved if a patient achieves either 1) a 30% increase in PD-1+ T cells in the peripheral blood in subjects who have a minimum of 25 cells/microliter (uL) 9 at baseline, or 2) an absolute increase of at least 75 PD-1+ T cells/uL in subjects who do not have a minimum of 25 PD-1+ T cells/uL at baseline.

SECONDARY OUTCOMES:
Safety including adverse events (AEs) and lab values | Up to 2 years post-enrollment.
  Grading of AEs and lab values will be according to Common Terminology Criteria for Adverse Events 5.0.
Overall response (OR) | Up to 5 years post-enrollment.
  OR will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hurwitz, MD, PhD, Principal Investigator — Yale University